CLINICAL TRIAL: NCT06805461
Title: A Multi-Center, Observational, Post-Marketing, Registry Study Following Patients With Solid Tumors Treated With Therapeutic Agents Via Localized Intra-Arterial Delivery Using the RenovoCath® Catheter
Brief Title: PanTheR Registry Trial
Acronym: PanTheR
Status: Recruiting | Type: Observational
Sponsor: RenovoRx (Industry)
Responsible Party: Sponsor
Other Study IDs: RR5
Record Dates: First submitted 2025-01-10; First posted 2025-02-03 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors
Keywords: Intra-Arterial Catheter

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients receiving Intra-Arterial treatment with RenovoCath: Patients receiving Intra-Arterial treatment with RenovoCath
  Interventions: Device: RenovoCath®

INTERVENTIONS:
Device: RenovoCath® — Intra-arterial catheter delivery of chemotherapy agents for the collection of real-world data.

SUMMARY:
This study is a multicenter, observational, post-marketing, registry study designed to track the safety and performance of the RenovoCath® device and assess survival outcomes in patients diagnosed with solid tumors who are treated with localized intra-arterial (IA) delivery of therapeutic agents to solid tumors using the RenovoCath® catheter.

DETAILED DESCRIPTION:
This study will enroll patients diagnosed with solid tumors who are willing to participate in the registry and meet the study enrollment criteria. Participants will be treated with therapeutic agents using RenovoCath® for the approved intended use according to the current country-specific Instructions for Use (IFU). Participants will be followed for survival outcome. Patients may chose to consent to participation in the registry before, during, or after treatment with the RenovoCath® device.

This observational post-marketing registry study is intended to track the safety and performance of the RenovoCath® device and assess patient survival / clinical outcomes of RenovoCath® in a real-world, clinical, observational setting when used for targeted delivery of therapeutic agents. Up to 1000 patients will be enrolled at up to an estimated 100 sites. Each patient participating in the registry study will have medical record retrievals including past data as of the time of their initial diagnosis through all localized IA administrations of therapeutic agent(s) using RenovoCath®, with continued record retrieval through the end of patient follow-up to record mortality rates. Patient data collection will include prior treatment history. Patients and/or their families will be contacted periodically after the treatment(s) to assess survival. It is anticipated that each participating patient's records will be retrieved approximately four times throughout the course of their treatment and follow-up, or retrospectively should patents decide to participate in the registry upon the completion of their treatment or during follow-up. This registry study is expected to continue for six years from study commencement.

ELIGIBILITY:
Eligibility Criteria:

1. Male and female patients who have been diagnosed with solid tumor cancers and are at least 18 years of age at the time of the first IA procedure
2. Patients willing to provide informed consent and HIPAA release for use of their relevant medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited for the study by treating physicians. Up to 1000 participants may be enrolled at up to an estimated 100 study sites. Participants will have been diagnosed with solid tumors with histological or cytological confirmation and may have been treated previously with chemotherapy, radiation therapy, or other modalities.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-09-03 (Estimated); Study Completion 2029-09-03 (Estimated)

PRIMARY OUTCOMES:
Safety of RenovoCath® as assessed by the number of participants experiencing adverse events related to the chemotherapy agents administered using RenovoCath. | From the time of the first treatment, until 30 days after the last treatment
  Number of participants experiencing adverse events related to the chemotherapy agents administered using RenovoCath.
Performance of RenovoCath® as assessed by the number of participants experiencing adverse events related to the inter-arterial drug delivery procedure. | From the time of the first treatment, until 30 days after the last treatment
  Track the performance of RenovoCath® in a real-world setting delivering a variety of therapeutic agents

SECONDARY OUTCOMES:
Overall Survival | 24 months from date of first treatment with IA
  Evaluate overall survival (OS) in patients diagnosed with solid tumors who undergo localized IA delivery of therapeutic agents via the RenovoCath®
Tumor Response Rate | 24 months from date of first treatment with IA
  Assess tumor response, via imaging, in the primary site of application
Number of participants who are downstaged and have their tumor resected after IA treatment with RenovoCth | 6 months from the date of the first IA treatment
  The number of participants who received IA treatment with RenovoCath and later receive resection of their tumor

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Baptist Health South Florida, Coral Gables, Florida
  - University of Pennsylvania Medical Center, Pittsburgh, Pennsylvania
  - The University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with participating investigators only.